CLINICAL TRIAL: NCT03700645
Title: Allopurinol in the Treatment of Patients With Diabetes Mellitus and Multivessel Coronary Artery Disease Treated by Either PCI or CABG: Pilot Study
Brief Title: Allopurinol in Diabetes Mellitus and Multivessel Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director. Research & development, Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-18-YA-354-18-CTIL
Record Dates: First submitted 2018-08-15; First posted 2018-10-09 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus; Ischemic Heart Disease; Multi Vessel Coronary Artery Disease
Keywords: Diabetes Mellitus; Uric asid; Multi Vessel Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus; Myocardial Ischemia | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PCI and standard medical treatment (No Intervention): Patients diagnosed with multi vessel disease that after Heart team discussion underwent intervention by PCI and receive standard medical treatment according to practice guidelines.
- PCI, standard treatment and Allopurinol (Active Comparator): Patients diagnosed with multi vessel disease that after Heart team discussion underwent intervention by PCI and in addition to standard medical treatment, receive treatment with allopurinol.
  Interventions: Drug: Allopurinol
- CABG and standard medical treatment (No Intervention): Patients diagnosed with multi vessel disease that after Heart team discussion underwent intervention by CABG and receive standard medical treatment according to practice guidelines.
- CABG standard treatment and Allopurinol (Active Comparator): Patients diagnosed with multi vessel disease that after Heart team discussion underwent intervention by CABG and in addition to standard medical treatment, receive treatment with allopurinol.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol
  Other Names: Alloril
  Arms: CABG standard treatment and Allopurinol; PCI, standard treatment and Allopurinol

SUMMARY:
Atherosclerosis is a progressive disease of the arterial wall, arising from the combination of endothelial dysfunction and inflammation. This link is exacerbated in diabetic patients.

Uric acid is known to generate oxidative stress and it's elevated levels has been shown to be associated with cardiac hypertrophy, inflammation, myocardial fibrosis and diastolic dysfunction. Allopurinol inhibits xanthine oxidase, an enzyme that regulates uric acid production. In observational studies it has been shown to reduce ischemia, inflammation and improve coronary flow. The aim of this study is to see whether treatment with Allopurinol in patients diagnosed with multivessel disease and undergoing treatment with either percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG) , will reduce markers of inflammation and improve quality of life and major adverse cardiovascular effects (MACE).

DETAILED DESCRIPTION:
This is a pilot study, PROBE design (prospective randomized open label blinded endpoints study), that will include 100 patients.

Patients will be recruited during their hospitalization in the cardiology department of Ichilov- Tel-Aviv Sourasky Medical Center.

It will include patients with known or newly diagnosed diabetes mellitus, hospitalized with diagnosis of acute coronary syndrome and multi-vessel coronary artery disease (CAD) that will be demonstrated by cardiac catheterization that the patients will undergo during their hospitalization in concordance with their diagnosis and practice guidelines.

The decision about intervention with either PCI or CABG will be accepted by a heart team after the initial demonstration of multi-vessel disease.

Study recruitment will take place either in the first 24 hours after PCI or before CABG.

All patients will sign an informed consent and randomized before any intervention is done.

After enrollment, patients will undergo the following baseline procedure (no later than 24 hours from PCI):

1. Physical examination and medical interview
2. Quality of life questionnaires (Seattle angina , EQ-5D)
3. Echocardiogram
4. Blood tests- see below for description
5. Endothelial function using the EndoPat®

Blood sampling will be done via IV cannula that will be placed in an antecubital vein. Blood sample analyses will be performed using reagents, calibrators and control materials in the local labs of each participating site. A 40 ml blood sample will be obtained for the following blood tests

1. Full chemistry including: lipid levels, thyroid function, liver enzymes function, Troponin, BNP, HbA1c, uric acid, creatinine and glucose levels.
2. Blood count
3. Inflammatory biomarker (hs-CRP, fibrinogen, IL-6, IL-1B, IL-18, MMP, IL-10, IL-35, TNFa, AchE , PAI-1, MPO, cholinergic status.)
4. Endothelial function markers: Endothelin-1, I-CAM, V-CAM, superoxide dismutase ADMA, and oxidized LDL
5. Oxidative Stress- superoxide dismutase ADMA, and oxidized LDL, Plasma protein carbonyls.
6. Urine samples- microalbuminuria, albumin/creatinine. Uric acid.

Endothelial function will be assessed using EndoPAT 2000 device (Itamar Medical Inc., Caesarea, Israel) that is a device that measures endothelial function using a sensor placed on the fingers. This device has been validated and used previously to assess peripheral arterial tone in other populations. EndoPAT bio-sensors are placed on the index fingers of both arms. EndoPAT quantifies the endothelium-mediated changes in vascular tone, elicited by a 5-minute occlusion of the brachial artery (using a standard blood pressure cuff). When the cuff is released, the surge of blood flow causes an endothelium-dependent Flow Mediated Dilatation (FMD). The dilatation, manifested as reactive hyperemia, is captured by EndoPAT as an increase in the PAT Signal amplitude. A post-occlusion to pre-occlusion ratio is calculated by the EndoPAT software, providing the EndoPAT index. In addition, the EndoPAT system will measure heart rate variability.

After randomization and assessment as described above, the patients will receive treatment according to the study arm they were assigned to which will include either standard medical therapy alone, or standard medical therapy and allopurinol.

Allopurinol will be given initially at 100 mg once daily dose, with dose escalation by 100 mg every 2 weeks till final dose of 300 mg daily will be reached.

After discharge, patients will be assessed several times:

1. One month after in cardiology clinic. Assessment will include all the tests as in the pre study exam (see above). also, patients will be monitored for the possible side effects of allopurinol treatment.
2. Three months- in cardiology clinic. Assessment will include all the tests as in the pre study exam (see above).

ELIGIBILITY:
Inclusion Criteria:

1. Acute Coronary Syndrome with positive troponin
2. Patients with known or newly diagnosed diabetes mellitus with HbA1c above 7% and below 10%
3. Patients above the age of 40
4. Stable Hemodynamic state (At least 12 hours from presentation with acute coronary syndrome)
5. Uric Acid > 6mg/dl or 355 micromol/l (males) and >5mg/dl or 297 Micromol/l (females)

Exclusion Criteria:

1. HbA1c below 7% or above 10%
2. Severe valvular insufficiency/Stenosis
3. Major surgery within 30 days
4. Any medical condition that would impair participation (e.g. progressive neurological disorders, mental illness)
5. Known intolerance/ current use of allopurinol/colchicine
6. Chronic inflammatory diseases: e.g. Lupus, rheumatoid arthritis, etc.
7. Current treatment with steroids, NSAID, chemotherapy or biologic medications
8. Extra-cardiac illness that is expected to limit survival to less than 2 years.
9. Past Cancer within the past 5 years (excluding BCC and SCC).

   -

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
hs-CRP | 3 months.
  Change in inflammatory biomarkers

SECONDARY OUTCOMES:
hs-CRP | one month
  Change in inflammatory biomarkers
Endothelial function markers | 3 month
  Endothelin-1, I-CAM, V-CAM, superoxide dismutase ADMA, and oxidized LDL, Change of RH-PAT
Heart rate variability | 3 month
  Heart rate variability
functional status and quality of life: the Seattle angina questionnaire | 3 month
  Quality of life evaluation- evaluates functional limitation in different activities due to chest pain and angina
Uric acid levels | one month and 3 month
  Uric acid levels
functional status, quality of life: EuroQol EQ-5D questionnaire | 3 month
  evaluation of degree of limitation in different daily activities
Reduction of peri-procedural myocardial infarction | 72 hours
  Reduction of peri-procedural myocardial infarction
MACE | 3 month
  major adverse cardiac events
Diastolic function | 3 month
  Diastolic function per echocardiogram- E/A
Diastolic function | 3 month
  Diastolic function per echocardiogram-E/E' med
Diastolic function | 3 month
  Diastolic function per echocardiogram- E/E' lat
Diastolic function | 3 month
  Diastolic function per echocardiogram- DT time

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Arbel, M.D, Principal Investigator — Tel Aviv University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Duckworth W, Abraira C, Moritz T, Reda D, Emanuele N, Reaven PD, Zieve FJ, Marks J, Davis SN, Hayward R, Warren SR, Goldman S, McCarren M, Vitek ME, Henderson WG, Huang GD; VADT Investigators. Glucose control and vascular complications in veterans with type 2 diabetes. N Engl J Med. 2009 Jan 8;360(2):129-39. doi: 10.1056/NEJMoa0808431. Epub 2008 Dec 17. PMID 19092145
- [Background] ACCORD Study Group; Gerstein HC, Miller ME, Genuth S, Ismail-Beigi F, Buse JB, Goff DC Jr, Probstfield JL, Cushman WC, Ginsberg HN, Bigger JT, Grimm RH Jr, Byington RP, Rosenberg YD, Friedewald WT. Long-term effects of intensive glucose lowering on cardiovascular outcomes. N Engl J Med. 2011 Mar 3;364(9):818-28. doi: 10.1056/NEJMoa1006524. PMID 21366473
- [Background] BARI 2D Study Group; Frye RL, August P, Brooks MM, Hardison RM, Kelsey SF, MacGregor JM, Orchard TJ, Chaitman BR, Genuth SM, Goldberg SH, Hlatky MA, Jones TL, Molitch ME, Nesto RW, Sako EY, Sobel BE. A randomized trial of therapies for type 2 diabetes and coronary artery disease. N Engl J Med. 2009 Jun 11;360(24):2503-15. doi: 10.1056/NEJMoa0805796. Epub 2009 Jun 7. PMID 19502645
- [Background] Look AHEAD Research Group; Wing RR, Bolin P, Brancati FL, Bray GA, Clark JM, Coday M, Crow RS, Curtis JM, Egan CM, Espeland MA, Evans M, Foreyt JP, Ghazarian S, Gregg EW, Harrison B, Hazuda HP, Hill JO, Horton ES, Hubbard VS, Jakicic JM, Jeffery RW, Johnson KC, Kahn SE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montez MG, Murillo A, Nathan DM, Patricio J, Peters A, Pi-Sunyer X, Pownall H, Reboussin D, Regensteiner JG, Rickman AD, Ryan DH, Safford M, Wadden TA, Wagenknecht LE, West DS, Williamson DF, Yanovski SZ. Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes. N Engl J Med. 2013 Jul 11;369(2):145-54. doi: 10.1056/NEJMoa1212914. Epub 2013 Jun 24. PMID 23796131
- [Background] Arbel Y, Zlotnik M, Halkin A, Havakuk O, Berliner S, Herz I, Rabinovich I, Keren G, Bazan S, Finkelstein A, Banai S. Admission glucose, fasting glucose, HbA1c levels and the SYNTAX score in non-diabetic patients undergoing coronary angiography. Clin Res Cardiol. 2014 Mar;103(3):223-7. doi: 10.1007/s00392-013-0641-7. Epub 2013 Nov 24. PMID 24271460
- [Background] de Mulder M, Umans VA, Cornel JH, van der Zant FM, Stam F, Oemrawsingh RM, Akkerhuis KM, Boersma E. Intensive glucose regulation in hyperglycemic acute coronary syndrome: results of the randomized BIOMarker study to identify the acute risk of a coronary syndrome-2 (BIOMArCS-2) glucose trial. JAMA Intern Med. 2013 Nov 11;173(20):1896-904. doi: 10.1001/jamainternmed.2013.10074. PMID 24018647
- [Background] Yang SW, Zhou YJ, Tian XF, Pan GZ, Liu YY, Zhang J, Guo ZF, Chen SY, Gao ST, Du J, Jia DA, Fang Z, Hu B, Han HY, Gao F, Hu DY, Xu YY; Beijing Heart and Metabolism Survey Study Group. Association of dysglycemia and all-cause mortality across the spectrum of coronary artery disease. Mayo Clin Proc. 2013 Sep;88(9):930-41. doi: 10.1016/j.mayocp.2013.05.022. PMID 24001485
- [Background] Neogi T, George J, Rekhraj S, Struthers AD, Choi H, Terkeltaub RA. Are either or both hyperuricemia and xanthine oxidase directly toxic to the vasculature? A critical appraisal. Arthritis Rheum. 2012 Feb;64(2):327-38. doi: 10.1002/art.33369. PMID 21953377
- [Background] Richette P, Perez-Ruiz F, Doherty M, Jansen TL, Nuki G, Pascual E, Punzi L, So AK, Bardin T. Improving cardiovascular and renal outcomes in gout: what should we target? Nat Rev Rheumatol. 2014 Nov;10(11):654-61. doi: 10.1038/nrrheum.2014.124. Epub 2014 Aug 19. PMID 25136785
- [Background] Jia G, Habibi J, Bostick BP, Ma L, DeMarco VG, Aroor AR, Hayden MR, Whaley-Connell AT, Sowers JR. Uric acid promotes left ventricular diastolic dysfunction in mice fed a Western diet. Hypertension. 2015 Mar;65(3):531-9. doi: 10.1161/HYPERTENSIONAHA.114.04737. Epub 2014 Dec 8. PMID 25489061
- [Background] Baena CP, Lotufo PA, Mill JG, Cunha Rde S, Bensenor IJ. Serum Uric Acid and Pulse Wave Velocity Among Healthy Adults: Baseline Data From the Brazilian Longitudinal Study of Adult Health (ELSA-Brasil). Am J Hypertens. 2015 Aug;28(8):966-70. doi: 10.1093/ajh/hpu298. Epub 2015 Jan 21. PMID 25609603
- [Background] Puddu P, Puddu GM, Cravero E, Vizioli L, Muscari A. Relationships among hyperuricemia, endothelial dysfunction and cardiovascular disease: molecular mechanisms and clinical implications. J Cardiol. 2012 May;59(3):235-42. doi: 10.1016/j.jjcc.2012.01.013. Epub 2012 Mar 6. PMID 22398104
- [Background] Gotsman I, Keren A, Lotan C, Zwas DR. Changes in uric acid levels and allopurinol use in chronic heart failure: association with improved survival. J Card Fail. 2012 Sep;18(9):694-701. doi: 10.1016/j.cardfail.2012.06.528. Epub 2012 Aug 3. PMID 22939038
- [Background] Miyaoka T, Mochizuki T, Takei T, Tsuchiya K, Nitta K. Serum uric acid levels and long-term outcomes in chronic kidney disease. Heart Vessels. 2014 Jul;29(4):504-12. doi: 10.1007/s00380-013-0396-0. Epub 2013 Aug 9. PMID 23929090
- [Background] Wu AH, Ghali JK, Neuberg GW, O'Connor CM, Carson PE, Levy WC. Uric acid level and allopurinol use as risk markers of mortality and morbidity in systolic heart failure. Am Heart J. 2010 Nov;160(5):928-33. doi: 10.1016/j.ahj.2010.08.006. PMID 21095282
- [Background] Ito H, Abe M, Mifune M, Oshikiri K, Antoku S, Takeuchi Y, Togane M. Hyperuricemia is independently associated with coronary heart disease and renal dysfunction in patients with type 2 diabetes mellitus. PLoS One. 2011;6(11):e27817. doi: 10.1371/journal.pone.0027817. Epub 2011 Nov 18. PMID 22125626
- [Background] Takagi H, Umemoto T. Atorvastatin therapy reduces serum uric acid levels: a meta-analysis of randomized controlled trials. Int J Cardiol. 2012 May 31;157(2):255-7. doi: 10.1016/j.ijcard.2012.01.092. Epub 2012 Feb 21. No abstract available. PMID 22360949
- [Background] Kanbay M, Segal M, Afsar B, Kang DH, Rodriguez-Iturbe B, Johnson RJ. The role of uric acid in the pathogenesis of human cardiovascular disease. Heart. 2013 Jun;99(11):759-66. doi: 10.1136/heartjnl-2012-302535. Epub 2013 Jan 23. PMID 23343689
- [Background] Fan Y, Wei F, Lang Y, Wang S. Losartan treatment for hypertensive patients with hyperuricaemia in Chinese population: a meta-analysis. J Hypertens. 2015 Apr;33(4):681-8; discussion 689. doi: 10.1097/HJH.0000000000000478. PMID 25915869
- [Background] El-Bassossy HM, Watson ML. Xanthine oxidase inhibition alleviates the cardiac complications of insulin resistance: effect on low grade inflammation and the angiotensin system. J Transl Med. 2015 Mar 6;13:82. doi: 10.1186/s12967-015-0445-9. PMID 25889404
- [Background] Erdogan D, Tayyar S, Uysal BA, Icli A, Karabacak M, Ozaydin M, Dogan A. Effects of allopurinol on coronary microvascular and left ventricular function in patients with idiopathic dilated cardiomyopathy. Can J Cardiol. 2012 Nov-Dec;28(6):721-7. doi: 10.1016/j.cjca.2012.04.005. Epub 2012 Jun 19. PMID 22717250
- [Background] Rekhraj S, Gandy SJ, Szwejkowski BR, Nadir MA, Noman A, Houston JG, Lang CC, George J, Struthers AD. High-dose allopurinol reduces left ventricular mass in patients with ischemic heart disease. J Am Coll Cardiol. 2013 Mar 5;61(9):926-32. doi: 10.1016/j.jacc.2012.09.066. PMID 23449426
- [Background] Thanassoulis G, Brophy JM, Richard H, Pilote L. Gout, allopurinol use, and heart failure outcomes. Arch Intern Med. 2010 Aug 9;170(15):1358-64. doi: 10.1001/archinternmed.2010.198. PMID 20696962
- [Background] de Abajo FJ, Gil MJ, Rodriguez A, Garcia-Poza P, Alvarez A, Bryant V, Garcia-Rodriguez LA. Allopurinol use and risk of non-fatal acute myocardial infarction. Heart. 2015 May;101(9):679-85. doi: 10.1136/heartjnl-2014-306670. Epub 2015 Jan 5. PMID 25561685
- [Background] Grimaldi-Bensouda L, Alperovitch A, Aubrun E, Danchin N, Rossignol M, Abenhaim L, Richette P; PGRx MI Group. Impact of allopurinol on risk of myocardial infarction. Ann Rheum Dis. 2015 May;74(5):836-42. doi: 10.1136/annrheumdis-2012-202972. Epub 2014 Jan 6. PMID 24395556
- [Background] Struthers A, Shearer F. Allopurinol: novel indications in cardiovascular disease. Heart. 2012 Nov;98(21):1543-5. doi: 10.1136/heartjnl-2012-302249. Epub 2012 Jul 16. No abstract available. PMID 22801998
- [Background] Rentoukas E, Tsarouhas K, Tsitsimpikou C, Lazaros G, Deftereos S, Vavetsi S. The prognostic impact of allopurinol in patients with acute myocardial infarction undergoing primary percutaneous coronary intervention. Int J Cardiol. 2010 Nov 19;145(2):257-258. doi: 10.1016/j.ijcard.2009.08.037. Epub 2009 Sep 22. PMID 19775763
- [Background] Givertz MM, Anstrom KJ, Redfield MM, Deswal A, Haddad H, Butler J, Tang WH, Dunlap ME, LeWinter MM, Mann DL, Felker GM, O'Connor CM, Goldsmith SR, Ofili EO, Saltzberg MT, Margulies KB, Cappola TP, Konstam MA, Semigran MJ, McNulty SE, Lee KL, Shah MR, Hernandez AF; NHLBI Heart Failure Clinical Research Network. Effects of Xanthine Oxidase Inhibition in Hyperuricemic Heart Failure Patients: The Xanthine Oxidase Inhibition for Hyperuricemic Heart Failure Patients (EXACT-HF) Study. Circulation. 2015 May 19;131(20):1763-71. doi: 10.1161/CIRCULATIONAHA.114.014536. Epub 2015 Apr 14. PMID 25986447
- [Background] Higgins P, Walters MR, Murray HM, McArthur K, McConnachie A, Lees KR, Dawson J. Allopurinol reduces brachial and central blood pressure, and carotid intima-media thickness progression after ischaemic stroke and transient ischaemic attack: a randomised controlled trial. Heart. 2014 Jul;100(14):1085-92. doi: 10.1136/heartjnl-2014-305683. Epub 2014 May 1. PMID 24790069
- [Background] Kao MP, Ang DS, Gandy SJ, Nadir MA, Houston JG, Lang CC, Struthers AD. Allopurinol benefits left ventricular mass and endothelial dysfunction in chronic kidney disease. J Am Soc Nephrol. 2011 Jul;22(7):1382-9. doi: 10.1681/ASN.2010111185. Epub 2011 Jun 30. PMID 21719783
- [Background] Erol T, Tekin A, Katircibasi MT, Sezgin N, Bilgi M, Tekin G, Zumrutdal A, Sezgin AT, Muderrisoglu H. Efficacy of allopurinol pretreatment for prevention of contrast-induced nephropathy: a randomized controlled trial. Int J Cardiol. 2013 Aug 20;167(4):1396-9. doi: 10.1016/j.ijcard.2012.04.068. Epub 2012 May 8. PMID 22572633
- [Background] Goicoechea M, Garcia de Vinuesa S, Verdalles U, Verde E, Macias N, Santos A, Perez de Jose A, Cedeno S, Linares T, Luno J. Allopurinol and progression of CKD and cardiovascular events: long-term follow-up of a randomized clinical trial. Am J Kidney Dis. 2015 Apr;65(4):543-9. doi: 10.1053/j.ajkd.2014.11.016. Epub 2015 Jan 13. PMID 25595565
- [Background] Noman A, Ang DS, Ogston S, Lang CC, Struthers AD. Effect of high-dose allopurinol on exercise in patients with chronic stable angina: a randomised, placebo controlled crossover trial. Lancet. 2010 Jun 19;375(9732):2161-7. doi: 10.1016/S0140-6736(10)60391-1. Epub 2010 Jun 9. PMID 20542554
- [Background] Guedes M, Esperanca A, Pereira AC, Rego C. What is the effect on cardiovascular events of reducing hyperuricemia with allopurinol? An evidence-based review. Rev Port Cardiol. 2014 Nov;33(11):727-32. doi: 10.1016/j.repc.2014.06.002. Epub 2014 Nov 20. English, Portuguese. PMID 25444231
- [Background] Castrejon I, Toledano E, Rosario MP, Loza E, Perez-Ruiz F, Carmona L. Safety of allopurinol compared with other urate-lowering drugs in patients with gout: a systematic review and meta-analysis. Rheumatol Int. 2015 Jul;35(7):1127-37. doi: 10.1007/s00296-014-3189-6. Epub 2014 Dec 18. PMID 25519877
- [Background] Kydd AS, Seth R, Buchbinder R, Falzon L, Edwards CJ, van der Heijde DM, Bombardier C. Urate-lowering therapy for the management of gout: a summary of 2 Cochrane reviews. J Rheumatol Suppl. 2014 Sep;92:33-41. doi: 10.3899/jrheum.140460. PMID 25180126
- [Background] Seth R, Kydd AS, Buchbinder R, Bombardier C, Edwards CJ. Allopurinol for chronic gout. Cochrane Database Syst Rev. 2014 Oct 14;2014(10):CD006077. doi: 10.1002/14651858.CD006077.pub3. PMID 25314636
- [Background] Spina M, Nagy Z, Ribera JM, Federico M, Aurer I, Jordan K, Borsaru G, Pristupa AS, Bosi A, Grosicki S, Glushko NL, Ristic D, Jakucs J, Montesinos P, Mayer J, Rego EM, Baldini S, Scartoni S, Capriati A, Maggi CA, Simonelli C; FLORENCE Study Group. FLORENCE: a randomized, double-blind, phase III pivotal study of febuxostat versus allopurinol for the prevention of tumor lysis syndrome (TLS) in patients with hematologic malignancies at intermediate to high TLS risk. Ann Oncol. 2015 Oct;26(10):2155-61. doi: 10.1093/annonc/mdv317. Epub 2015 Jul 27. PMID 26216382